CLINICAL TRIAL: NCT01631565
Title: Management of Symptoms in Patients With Advanced Lung Cancer: Early Incorporation of Patient and Family to Attention and Care Program in Oncology
Brief Title: Early Incorporation of Patient and Family to Attention and Care Program in Oncology Versus Standard of Care
Acronym: PACO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez MD, SNI II, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PACO2012
Record Dates: First submitted 2012-06-11; First posted 2012-06-29 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Lung Neoplasms
Keywords: Palliative Care; Survival; Quality of life
MeSH Terms: conditions — Lung Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (No Intervention): Usual care given to the patients. Treatment, follow-up.
- Early Palliative Care (Experimental): Intervention: Early allocation to palliative care. Intervention: Nutritional counseling. Intervention: patient and care-taker psychoeducation, depression and anxiety evaluation.
  Standard of care: Oncological treatment according to stage of disease (IIIb/IV).
  Treatment: Chemotherapy (platins, taxans, TKIs) Baseline: BMI, and anthropometric characteristics (weight, height). Follow-up: During 6 chemotherapy circles with: Quality of Life (EORTC qlq-c30), HADS, ESAS and ZARIT.
  Interventions: Behavioral: Early allocation to palliative care; Behavioral: Nutritional counseling; Behavioral: Psychoeducation.

INTERVENTIONS:
Behavioral: Early allocation to palliative care — Symptoms management (e.g. Pain, nausea, dehydration management).
  Other Names: experimental
  Arms: Early Palliative Care
Behavioral: Nutritional counseling — Nutritional status evaluation and dietary supplementation according to the patient requirements.
  Arms: Early Palliative Care
Behavioral: Psychoeducation. — Patient and care-taker psychoeducation, depression and anxiety evaluation.
  Arms: Early Palliative Care

SUMMARY:
There is recent evidence that early palliative care administered to patients helps for their quality of life (QoL). It is however not part of the standard multidisciplinary treatment.

This study intents to evaluate the effect of early palliative care in patients with advanced Non-Small Cell Lung Cancer (NSCLC) compared to the standard of care.

DETAILED DESCRIPTION:
The multidisciplinary approach of palliative care for symptom management has an impact on the quality of life (QoL) of patients and their families. The World Health Organization (WHO) and the American Society of Clinical Oncology (ASCO) recommend incorporating early palliative care, simultaneously with cancer treatment. Unfortunately, this recommendation has not been followed in many cancer centers and late referrals to hospice are still frequent.

Patients with lung cancer have more symptoms than patients with other cancer. The impact on QoL and symptom management has acquired a great relevance. However, few studies demonstrating the benefit of early incorporation of palliative care in the management of patients with advanced lung cancer have been shown.

Palliative care is defined as the care given to patients with progressive active and advanced disease, and its main purpose is the relief and prevention of suffering and improving QoL.

In Mexico, the law defines palliative care as comprehensive care for those illnesses not responsive to curative treatment and include, but are not limited, to pain and other symptoms associated with the disease and psychological care, social and spiritual, of the patients and their families.

Psychological aspects The psychological manifestations in patients with lung cancer are determined by several factors. Depression and anxiety are the most common psychological reactions. It has been identified that 25% of cancer patients suffer from major depression at some point during the course of the disease and has been associated with decreased survival and QoL. Patients with anxiety disorders become more attached to medical treatment but seek alternative treatments more often. The main objective of psychological interventions is reducing maladaptive emotional reactions. In advanced stages, caregivers also confront stress and depression that could lead to health problems.

Nutritional aspects Malnutrition is reported in 60 to 79% in patients with lung cancer and is the largest contribution to morbidity and mortality. Cachexia is responsible directly or indirectly to death in one third of patients. The objectives of nutritional support are: improving tolerance to specific cancer treatment, decreasing the incidence of complications and, improving the QoL. Thus, it is necessary to conduct an early diagnosis of nutritional status in order to design nutritional intervention and improve their sense of comfort and QoL.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage IV
* ECOG 0-2
* Patients treated virgin
* Receive platinum-based chemotherapy

Exclusion Criteria:

* Suicide Risk
* Delirium
* Cognitive impairment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Global survival | from inclusion until at least 6 months after
  Overall survival will be determined from the date of commencement of treatment to date of death, regardless of the cause of death. In patients who did not die at the time of final analysis will use the date of last contact.

SECONDARY OUTCOMES:
Progression Free Survival | from inclusion until at least 6 months after
  Is defined as the time from start of treatment until the date of the first documented evidence of progression (RECIST criteria) or the date of death for any reason in the absence of disease progression (EP). For patients who have died or progressed at the time of final analysis, use the date of last contact.
Quality of life | from inclusion until at least 6 months after
  by EORTC QLQ C30, QLQ LC13

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta, MD Msc, Principal Investigator — Mexico. Nacional Cancer Institute
Locations (1):
- National Cancer Institute- México, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gore JM, Brophy CJ, Greenstone MA. How well do we care for patients with end stage chronic obstructive pulmonary disease (COPD)? A comparison of palliative care and quality of life in COPD and lung cancer. Thorax. 2000 Dec;55(12):1000-6. doi: 10.1136/thorax.55.12.1000. PMID 11083884
- [Background] Nieder C, Norum J. Early palliative care in patients with metastatic non-small cell lung cancer. Ann Palliat Med. 2012 Apr;1(1):84-6. doi: 10.3978/j.issn.2224-5820.2012.03.05. No abstract available. PMID 25841435
- [Background] Follwell M, Burman D, Le LW, Wakimoto K, Seccareccia D, Bryson J, Rodin G, Zimmermann C. Phase II study of an outpatient palliative care intervention in patients with metastatic cancer. J Clin Oncol. 2009 Jan 10;27(2):206-13. doi: 10.1200/JCO.2008.17.7568. Epub 2008 Dec 8. PMID 19064979
- [Background] Jordhoy MS, Fayers P, Loge JH, Ahlner-Elmqvist M, Kaasa S. Quality of life in palliative cancer care: results from a cluster randomized trial. J Clin Oncol. 2001 Sep 15;19(18):3884-94. doi: 10.1200/JCO.2001.19.18.3884. PMID 11559726
- [Background] Ferris FD, Bruera E, Cherny N, Cummings C, Currow D, Dudgeon D, Janjan N, Strasser F, von Gunten CF, Von Roenn JH. Palliative cancer care a decade later: accomplishments, the need, next steps -- from the American Society of Clinical Oncology. J Clin Oncol. 2009 Jun 20;27(18):3052-8. doi: 10.1200/JCO.2008.20.1558. Epub 2009 May 18. PMID 19451437
- [Background] Akechi T, Okuyama T, Akizuki N, Azuma H, Sagawa R, Furukawa TA, Uchitomi Y. Course of psychological distress and its predictors in advanced non-small cell lung cancer patients. Psychooncology. 2006 Jun;15(6):463-73. doi: 10.1002/pon.975. PMID 16173112
- [Derived] Allende S, Turcott JG, Verastegui E, Rodriguez-Mayoral O, Flores-Estrada D, Perez Camargo DA, Ramos-Ramirez M, Martinez-Hernandez JN, Onate-Ocana LF, Pina PS, Cardona AF, Arrieta O. Early Incorporation to Palliative Care (EPC) in Patients With Advanced Non-Small Cell Lung Cancer: The PACO Randomized Clinical Trial. Oncologist. 2024 Oct 3;29(10):e1373-e1385. doi: 10.1093/oncolo/oyae050. PMID 38558247